CLINICAL TRIAL: NCT05118958
Title: A Multiple Part, Phase 1 Crossover Study in Healthy Subjects to Evaluate the Pharmacokinetic (PK) Profile of KVD824 Following Single and Multiple Doses of Novel KVD824 Modified Release (MR) Formulations Compared to a Reference KVD824 Immediate Release (IR) Formulation
Brief Title: Phase 1 Crossover Study in Healthy Subjects to Evaluate the PK Profile of KVD824 Following Single and Multiple Doses of Modified Release (MR) Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KVD824-102
Record Dates: First submitted 2021-10-26; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Initial open-label crossover (Part 1) followed by double-blind, randomised, placebo-controlled part (Part 3).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part 1 - Period 1 - Prototype 1 600 mg (single dose fasted) (Experimental): 600 mg (2 x 300 mg) KVD824 prototype 1 modified-release tablet dosed orally in fasted state as a single dose
  Interventions: Drug: KVD824 Prototype 1 modified-release tablet
- Part 1 - Period 3 - Prototype 2 600 mg (single dose fasted) (Experimental): 600 mg (2 x 300 mg) KVD824 prototype 2 modified-release tablet dosed orally in fasted state as a single dose
  Interventions: Drug: KVD824 Prototype 2 modified-release tablet
- Part 1 - Period 4 - Prototype 1 900 mg (single dose fasted) (Experimental): 900 mg (3 x 300 mg) KVD824 prototype 1 modified-release tablet dosed orally in fasted state as a single dose
  Interventions: Drug: KVD824 Prototype 1 modified-release tablet
- Part 1 - Period 5 - Prototype 1 600 mg and Prototype 3 300 mg (single dose fasted) (Experimental): 600 mg (2 x 300 mg) KVD824 prototype 1 modified-release tablet plus 300 mg (1 x 300 mg) Prototype 3 dosed orally in fasted state as a single dose
  Interventions: Drug: KVD824 Prototype 1 modified-release tablet; Drug: KVD824 Prototype 3 modified-release tablet
- Part 1 - Period 6 - Prototype 1 900 mg (single dose fed) (Experimental): 900 mg (3 x 300 mg) KVD824 prototype 1 modified-release tablet dosed orally in fed state as a single dose
  Interventions: Drug: KVD824 Prototype 1 modified-release tablet
- Part 3 - KVD824 Prototype 1 600 mg (multiple dose fed) (Experimental): 600 mg (2 x 300 mg) KVD824 prototype 1 modified-release tablet dosed orally twice daily in fed state for 13 days with a single dose on day 14.
  Interventions: Drug: KVD824 Prototype 1 modified-release tablet
- Part 3 - Placebo to KVD824 Prototype 1 600 mg (multiple dose fed) (Placebo Comparator): Placebo to 600 mg KVD824 prototype 1 modified-release tablet dosed orally twice daily in fed state for 13 days with a single dose on day 14.
  Interventions: Drug: Placebo to KVD824 Prototype 1
- Part 3 - KVD824 Prototype 1 900 mg (multiple dose fed) (Experimental): 900 mg (3 x 300 mg) KVD824 prototype 1 modified-release tablet dosed orally twice daily in fed state for 13 days with a single dose on day 14.
  Interventions: Drug: KVD824 Prototype 1 modified-release tablet
- Part 3 - Placebo to KVD824 Prototype 1 900 mg (multiple dose fed) (Placebo Comparator): Placebo to 900 mg KVD824 prototype 1 modified-release tablet dosed orally twice daily in fed state for 13 days with a single dose on day 14.
  Interventions: Drug: Placebo to KVD824 Prototype 1
- Part 3 - KVD824 Prototype 1 900 mg (multiple dose fasted) (Experimental): 900 mg (3 x 300 mg) KVD824 prototype 1 modified-release tablet dosed orally twice daily in fasted state for 13 days with a single dose on day 14.
  Interventions: Drug: KVD824 Prototype 1 modified-release tablet
- Part 3 - Placebo to KVD824 Prototype 1 900 mg (multiple dose fasted) (Placebo Comparator): Placebo to 900 mg KVD824 prototype 1 modified-release tablet dosed orally twice daily in fasted state for 13 days with a single dose on day 14.
  Interventions: Drug: Placebo to KVD824 Prototype 1
- Part 1 - Period 2 - KVD824 IR Capsule 600 mg (single dose fasted) (Active Comparator): 600 mg (2 x 300 mg) KVD824 immediate release Capsule dosed orally in fasted state as a single dose
  Interventions: Drug: KVD824 Immediate-Release Capsule

INTERVENTIONS:
Drug: KVD824 Prototype 1 modified-release tablet — 300 mg modified-release tablet
  Arms: Part 1 - Period 1 - Prototype 1 600 mg (single dose fasted); Part 1 - Period 4 - Prototype 1 900 mg (single dose fasted); Part 1 - Period 5 - Prototype 1 600 mg and Prototype 3 300 mg (single dose fasted); Part 1 - Period 6 - Prototype 1 900 mg (single dose fed); Part 3 - KVD824 Prototype 1 600 mg (multiple dose fed); Part 3 - KVD824 Prototype 1 900 mg (multiple dose fasted); Part 3 - KVD824 Prototype 1 900 mg (multiple dose fed)
Drug: KVD824 Prototype 2 modified-release tablet — 300 mg modified-release tablet
  Arms: Part 1 - Period 3 - Prototype 2 600 mg (single dose fasted)
Drug: KVD824 Immediate-Release Capsule — 300 mg immediate-release capsule
  Arms: Part 1 - Period 2 - KVD824 IR Capsule 600 mg (single dose fasted)
Drug: Placebo to KVD824 Prototype 1 — Placebo to 300 mg KVD824 Prototype 1 modified-release tablet
  Arms: Part 3 - Placebo to KVD824 Prototype 1 600 mg (multiple dose fed); Part 3 - Placebo to KVD824 Prototype 1 900 mg (multiple dose fasted); Part 3 - Placebo to KVD824 Prototype 1 900 mg (multiple dose fed)
Drug: KVD824 Prototype 3 modified-release tablet — 300 mg modified-release tablet
  Arms: Part 1 - Period 5 - Prototype 1 600 mg and Prototype 3 300 mg (single dose fasted)

SUMMARY:
This is a 3 part, phase 1 crossover study in healthy subjects to evaluate the pharmacokinetic profile of KVD824 following single and multiple doses of novel KVD824 modified-release formulations compared with a reference KVD824 immediate release formulation.

DETAILED DESCRIPTION:
Part 1 of the study was a single-centre, open-label, non-randomised, 6-period crossover study designed to investigate the PK and safety of KVD824 MR prototype formulations (with or without an additional KVD824 IR capsule) compared to a reference KVD824 IR capsule formulation in healthy male and female subjects. Part 2 was an optional part designed to investigate the PK and safety of a selected KVD824 MR prototype tablet formulation (with or without an additional KVD824 IR capsule) in healthy male and female subjects in both the fed and fasted state. Note: this Part was not conducted as sufficient information on food effect was collected in the other Parts of the study.

Part 3 was a single-centre, randomised, double-blind, placebo-controlled, multiple dose group study to investigate the PK and safety of a selected KVD824 MR prototype tablet formulation (with or without an additional KVD824 IR capsule) in healthy male and female subjects. Part 3 started following completion of Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females.
2. Aged 18 to 55 years, inclusive at the time of signing informed consent.
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening.
4. Must be willing and able to communicate and participate in the whole study.
5. Must provide written informed consent.
6. Must agree to adhere to the contraception requirements.

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1.
2. Subjects who are study site employees, sponsor employees, or immediate family members of site or sponsor employees.
3. Subjects who have previously been administered IMP in this study. Subjects who have taken part in one part of this study are not permitted to take part in any other study part.
4. History of any drug or alcohol abuse in the past 2 years.
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type).
6. A confirmed positive alcohol breath test at screening or admission.
7. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
9. Females of childbearing potential who are pregnant or lactating (all female subjects must have a negative serum pregnancy test at screening and urine pregnancy test on admission).
10. Subjects with pregnant or lactating partners.
11. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening.
12. Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are allowed.
13. Confirmed positive drugs of abuse test result.
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
15. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <70 mL/min using the Cockcroft-Gault equation.
16. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator.
17. Subjects with a history of cholecystectomy or gall stones.
18. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
19. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
20. Donation or loss of greater than 400 mL of blood within the previous 3 months.
21. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day, HRT or hormonal contraception) in the 14 days before IMP administration.
22. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Tlag | Days 1, 10 and 14
  Time prior to the first measurable concentration after single and multiple doses of KVD824
Pharmacokinetics - Tmax | Days 1, 10 and 14
  Time of maximum observed concentration after single and multiple doses of KVD824 with and without food
Pharmacokinetics - Cmax | Days 1, 10 and 14
  Maximum observed concentration after single and multiple doses of KVD824 with and without food
Pharmacokinetics - Cmax/Dose | Days 1, 10 and 14
  Maximum observed concentration divided by dose
Pharmacokinetics - C12 | Days 1, 10 and 14
  Plasma concentration observed at time 12 h after single and multiple doses
Pharmacokinetics - C24 | Days 1, 10 and 14
  Plasma concentration observed at time 24 h after single and multiple doses
Pharmacokinetics - Ctrough | Days 2-14
  Concentration prior to the morning dose on Days 2-14 and prior to the evening dose on Days 2-13
Pharmacokinetics - Cmin | Days 2-14
  Minimum observed concentration during the dosing interval (between dose time and dose time plus tau) after single and multiple doses of KVD824 with and without food
Pharmacokinetics - Cavg | Days 2-14
  Average concentration (AUC(0-tau)/tau)
Pharmacokinetics - AUC(0-12) | Days 1, 10 and 14
  Area under the curve from time 0 to 12 hours post-dose after single and multiple doses
Pharmacokinetics - AUC(0-12)/Dose | Days 1, 10 and 14
  Area under the curve from time 0 to 12 hours post-dose divided by dose
Pharmacokinetics - AUC(0-24) | Days 1, 10 and 14
  Area under the curve from time 0 to 24 hours post-dose after single and multiple doses
Pharmacokinetics - AUC(0-24)/Dose | Days 1, 10 and 14
  Area under the curve from time 0 to 24 hours post-dose divided by dose
Pharmacokinetics - AUC(0-last) | Days 1, 10 and 14
  Area under the curve from time 0 to the time of last measurable concentration after single and multiple doses
Pharmacokinetics - AUC(0-last)/Dose | Days 1, 10 and 14
  Area under the curve from time 0 to the time of last measurable concentration divided by dose
Pharmacokinetics - AUC(0-tau) | Days 1, 10 and 14
  Area under the curve for the defined interval between doses (tau)
Pharmacokinetics - AUC(0-inf) | Days 1, 10 and 14
  Area under the curve from time 0 extrapolated to infinity
Pharmacokinetics - AUC(0-inf)/D | Days 1, 10 and 14
  Area under the curve from time 0 extrapolated to infinity divided by dose
Pharmacokinetics - AUCextrap | Days 1, 10 and 14
  Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity
Pharmacokinetics - T1/2 | Days 1, 10 and 14
  Terminal elimination half-life after single and multiple doses of KVD824 with and without food
Pharmacokinetics - Lambda-z | Days 1, 10 and 14
  First order rate constant associated with the terminal (log-linear) portion of the curve after single and multiple doses
Pharmacokinetics - CL/F | Days 1, 10 and 14
  Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown
Pharmacokinetics - CL/Ftau | Days 1, 10 and 14
  Total body clearance calculated using AUC(0-tau) after repeated extravascular administration, where F (fraction of dose bioavailable) is unknown
Pharmacokinetics - Vz/F | Days 1, 10 and 14
  Apparent volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown
Pharmacokinetics - Vz/Flau | Days 1, 10 and 14
  Apparent volume of distribution based on the terminal phase calculated using AUC(0-tau) after extravascular administration where F (fraction of dose bioavailable) is unknown
Pharmacokinetics - Frel Cmax | Days 1, 10 and 14
  Relative bioavailability based on Cmax
Pharmacokinetics - Frel AUC(0-12) | Days 1, 10 and 14
  Relative bioavailability based on AUC(0-12)
Pharmacokinetics - Frel AUC(0-inf) | Days 1, 10 and 14
  Relative bioavailability based on AUC(0-inf)
Pharmacokinetics - AR Cmax | Days 1, 10 and 14
  Accumulation ratio based on Cmax repeated dose/Cmax single dose
Pharmacokinetics - Fluctuation | Days 1, 10 and 14
  Peak to trough fluctuation (Cmax-Cmin)/Cavg × 100

SECONDARY OUTCOMES:
Safety - Adverse Events | Change from pre-dose to last visit (up to 14 days)
  Number of Subjects with Adverse Events
Safety - Serious Adverse Events | Change from pre-dose to last visit (up to 14 days)
  Number of Subjects with Serious Adverse Events
Safety - Laboratory Assessments | Throughout the trial to last visit (up to 14 days)
  Number of participants with clinically significant changes in laboratory assessments
Safety - Vital Signs | Throughout the trial to last visit (up to 14 days)
  Number of participants with clinically significant changes in vital signs
Safety - ECG | Throughout the trial to last visit (up to 14 days)
  Number of participants with clinically significant changes in electrocardiogram (ECG) measurements

CONTACTS AND LOCATIONS:
Locations (1):
- KalVista Investigative Site, Nottingham, United Kingdom